CLINICAL TRIAL: NCT00345904
Title: A Phase III Study for Evaluation of Immunogenicity and Reactogenicity of Fluarix™ (Influsplit SSW®) 2006/2007 in People Aged 18 Years or Above
Brief Title: Study to Evaluate the Safety and Immunogenicity of Fluarix™ 2006/2007 in Adults Aged 18 Years or Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 107507
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Influenza
Keywords: influenza, vaccine; prophylaxis of influenza
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

INTERVENTIONS:
Biological: Fluarix

SUMMARY:
Vaccination is currently the most effective mean of controlling influenza and preventing its complications and mortality in persons at risk. Because of the variable nature of influenza viruses, the composition of influenza vaccines changes almost every year, to target the 3 main circulating strains. Each year the influenza vaccine formulation may thus be different and clinical studies are mandated to ensure that the immunogenicity and safety of the vaccine formulated from the three annual circulating strains are similar to what was observed during the previous years.

This study is designed to test the immunogenicity and reactogenicity of the Fluarix™ vaccine containing the influenza strains recommended for the 2006-2007 season.

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged 18 years or above at the time of the vaccination;
* Healthy subjects or with well-controlled chronic diseases;
* If the subject is female, she must be of non-childbearing potential

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the vaccination or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned during the study.
* Administration of an influenza vaccine within 6 months preceding the study start.
* Administration of an influenza vaccine other than the study vaccine during the entire study
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Not stabilized or clinically serious chronic underlying disease
* Lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-07; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
to evaluate the humoral immune response in terms of anti-Haemmagglutinin antibodies 21 days post-vaccination

SECONDARY OUTCOMES:
To evaluate the safety and reactogenicity of the vaccine in term of solicited local and general adverse events, unsolicited adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Germany (2):
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 107507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register